CLINICAL TRIAL: NCT01269632
Title: Long Term Evaluation of Young Adults Born to HIV-infected Mothers. A Cohort of Young Adults Infected With HIV Since Birth or During Childhood
Brief Title: Cohort of Young Adults Infected With HIV Since Birth or During Childhood
Acronym: CO19 COVERTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2009-AO1219-48
Record Dates: First submitted 2010-09-17; First posted 2011-01-04 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2018-07

CONDITIONS: HIV Infection; Young Adult
Keywords: teenagers to adult transition; comparison
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection; Biological Specimen Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV infected (Other): young adult infected by HIV
  Interventions: Biological: blood sampling, specific biological exams and biobank and self administered questionnaires
- HIV uninfected (Other): a control group of HIV uninfected young adult will be included for comparison in physiopathological module (metabolic, cardiovascular, and immunological)
  Interventions: Biological: blood sampling, specific biological exams and biobank and self administered questionnaires

INTERVENTIONS:
Biological: blood sampling, specific biological exams and biobank and self administered questionnaires — HIV INFECTION at inclusion and annually up to 06 years follow-up
  1. clinical and therapeutic evaluation by physician
  2. biological: blood sampling, specific biological exams and biobank
  3. self administered questionnaires
  In the physiopathological module: at inclusion and after 3 years follow up: OGTT, CT Scan, Dexa Scan, cardiovascular explorations (carotid intima media thickness, pulse wave velocity, transthoracic echocardiography)
  HIV UNINFECTED at inclusion and after 3 years follow up
  1. clinical evaluation by physician
  2. biological: blood sampling, specific biological exams and biobank
  3. self administered questionnaires

SUMMARY:
Background: With the improvement of the prognosis for HIV-infected infants, thanks to the availability of antiretroviral therapies, young adults infected with HIV since birth are becoming an emerging group among the HIV-infected population. Morbidity, mortality and immunovirological evolution in these young adults need to be studied in a large population and compared to patients infected with HIV later in adulthood or to the general population in terms of mortality. Moreover, the study of accelerated or premature ageing, linked to HIV and/or antiretroviral therapy, is particularly interesting in this population.

Objectives: To study the transition to adulthood and the further evolution of HIV-1 or -2 perinatally infected young adults: 1) To study the teenager to adult transition in terms of clinical and immunovirological status, schooling and professional integration, sexuality and reproductive life, transition from paediatrics to adult departments; 2) To study prognosis, morbidity and mortality according to age, infection stage at the time of antiretroviral initiation and therapeutic history; 3) To study the incidence and expression of adverse events and the potential link to antiretroviral therapies; 4) To study the markers of a potential premature ageing, from the metabolic, cardiovascular and immunological points of view.

DETAILED DESCRIPTION:
Methods: A national multicenter cohort of young adults, infected with HIV since birth or during childhood, including a common module and a physiopathological module (metabolic,, cardiovascular and immunological). A control group of HIV-uninfected young adults is included for comparison in the latter module. Patients aged between 18 and 25 years of age, whose HIV diagnosis was made before the age of 13 are eligible for ANRS CO19 COVERTE. This cohort is an extension of the EPF cohort (ANRS CO10), in which follow-up stops at the age 18, with an extension to adults with a HIV diagnosis established before the age of 13. Questionnaires are filled out by physicians once a year. Self-administered questionnaires are also carried out. Blood sampling and specific biological exams are collected and a biobank constituted. In the physiopathological module, specific exams are carried out at inclusion and after 3 years of follow-up: metabolic and immunological exams, OGTT, CT-scan and DXA-scan, and cardiovascular explorations (carotid intima-media thickness, pulse wave velocity …). An estimated 400 enrolments during the first 3 years is expected in the common module and an estimated 200 HIV-infected subjects and 75 uninfected controls is expected in the physiopathological module.

Expected results: The follow-up of young adults in this cohort will bring new data on the long term efficacy of antiretroviral treatment and their adverse events, from the metabolic, cardiovascular and immunological, point of view, be they linked or not to HIV infection per se. This analysis will take into account the characteristics of this population, as compared to adults infected during adulthood: an early exposure to HIV and antiretroviral treatment, a different social context, difficulties in care, and a different exposure to risk factors for adverse events and complications. We will evaluate the impact of the transition to adulthood and of the transition from paediatrics to adult departments, on clinical prognosis, adherence, professional and schooling integration, sexuality, social life.

ELIGIBILITY:
Group of HIV Infection

Inclusion Criteria:

* Age ≥ 18 and < 25 years
* Able to give written consent
* Covered by French Social Security
* diagnosis of HIV-1 et/ou-2 documented before age 13

Exclusion Criteria (for physiopathological module only)

* Under protection(saving) of justice

Control Group

Inclusion Criteria:

* Age ≥ 18 and ≤ 25 years
* Able to give written consent
* Covered by French Social Security
* With a brother or sister, cousin, father or mother HIV infected, inbred or adopted
* With a negative serology for HIV infection, HBV, HCV
* Without diabetes mellitus
* able to go to Clinical Investigation Center of Necker and to Hospital St. Antoine for the recruitment and monitoring

Exclusion Criteria:

* Under protection(saving) of justice

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 469 (Actual)
Dates: Start 2010-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Immuno virological and clinical prognosis: HIV RNA <50c/mL, CD4 cells count>500 cells/mL, vital status, CDC stage | at inclusion and annually up to 06 years follow-up

SECONDARY OUTCOMES:
Professional and schooling integration, social life:marital status, type of accommodation, education level, type and age at first employment | at inclusion and annually up to 6 years follow up
sexuality, sexual risk behaviour: age at first intercourse, condom use at first, last sexual intercourse, and during last year, unplanned pregnancy, interruption of pregnancy | at inclusion and annually up to 6 year follow-up
metabolic and cardiovascular abnormalities: abnormalities in glucose tolerance and insulino-resistance, dyslipidemia, lipodystrophy, adipocyte dysfunction, atherosclerosis,dysfunction, median of intima media thickness and pulse wave velocity | at inclusion and after 3 years follow-up
Lymphocyte phenotype and functional capacity of T lymphocyte: description of dysfunctional CMV-specific T cell, T cell responses measured at inclusion, and their evolution during follow-up | at inclusion and after 3 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hugues Aumaitre, Principal Investigator — Centre hospitalier de Perpignan; Eric Froguel, Principal Investigator — Hopital de Lagny; Michèle Bentata, Principal Investigator — Hopital Avicenne; Philippe Genet, Principal Investigator — Hopital Argenteuil; Olivier Patey, Principal Investigator — CHIC Villeneuve St Georges; Laurence Gerard, Principal Investigator — St Louis Paris; Frédéric Lucht, Principal Investigator — St Etienne; Bruno Hoen, Principal Investigator — St Jacques Besançon; Jean Luc Schmit, Principal Investigator — Hôpital Nord Amiens; Claire Pintado, Principal Investigator — St Louis Paris; Cécile Goujard, Principal Investigator — Le Kremlin Bicetre; Thierry Allegre, Principal Investigator — CH Aix en Provence; Alain Lafeuillade, Principal Investigator — CHIC Toulon; Pierre De Truchis, Principal Investigator — Raymond Poincarré Garches; Vincent Jeantils, Principal Investigator — Jean Verdier Bondy; Claudine Duvivier, Principal Investigator — Institut Pasteur; Laurence Slama, Principal Investigator — Tenon Paris; Olivier Bouchaud, Principal Investigator — Hopital Avicenne Bobigny; Marie Karmochkine, Principal Investigator — Georges Pompidou Paris; Dominique Salmon Ceron, Principal Investigator — Cochin Paris; Emmanuel Mortier, Principal Investigator — Louis Mourier Colombes; Roland Tubiana, Principal Investigator — Pitié Salpétrière Paris; Pierre Marie Girard, Principal Investigator — St Antoine Paris; André Cabié, Principal Investigator — CHU Fort de France; Jean Marie Chennebault, Principal Investigator — University Hospital, Angers; Philippe Morlat, Principal Investigator — St André Bordeaux; Pierre Weinbreck, Principal Investigator — Hôpital Dupuytren; Laurent Cotte, Principal Investigator — La Croix Rousse Lyon; Sophie Matheron, Principal Investigator — Bichat Paris; Véronique Reliquet, Principal Investigator — Hotel Dieu Nantes; Philippe Pérré, Principal Investigator — CHD Les Oudairies La Roche Sur Yon; Cédric Arvieux, Principal Investigator — Hopital Pontchaillou Rennes; Christine Cheneau, Principal Investigator — Centre Hospitalier Strasbourg; Martine Obadia, Principal Investigator — CH Purpan Toulouse; Renaud Verdon, Principal Investigator — CHU Cote de Nacre Caen; Christine Jacomet, Principal Investigator — Hopital Gabriel Montpied Clermont Ferrand; Lionel Piroth, Principal Investigator — CHU Hopital d'enfants Dijon; Antoine Chéret, Principal Investigator — CH TOURCOING; Yasmine Debab, Principal Investigator — CHU Charles Nicolle Rouen; Dominique Merrien, Principal Investigator — CH Compiègne; Patrick Mercié, Principal Investigator — CHU St André Bordeaux; Valérie Garrait, Principal Investigator — CHIC Créteil; Marie Aude Khuong, Principal Investigator — Centre Hospitalier Général St Denis; Geneviève Beck Wirth, Principal Investigator — CH Mulhouse; Stéphane Blanche, Principal Investigator — Necker Paris; Franck Boccara, Principal Investigator — St Antoine Paris; Claudine Barbuat, Principal Investigator — CHR Caremeau Nimes; Jean Paul Viard, Principal Investigator — Hotel Dieu Paris; Ghislaine Firtion, Principal Investigator — Cochin Paris; Albert Faye, Principal Investigator — Robert Debré Paris; Catherine Dollfus, Principal Investigator — Armand Trousseau Paris; Corinne Floch Tudal, Principal Investigator — Louis Mourier Colombes; Kamila Kebaili, Principal Investigator — Hopital de jour ISHOP Lyon; Joelle Tricoire, Principal Investigator — CHU Paule de Viguier Toulouse; Françoise Mazingue, Principal Investigator — CHR Jeanne de Flandres Lille; Pascal Bolot, Principal Investigator — CHG St Denis; Francois Bissuel, Principal Investigator — CH LC Fleming St Martin Guadeloupe; Anne Chace, Principal Investigator — CHIC Villeneuve St Georges; Narcisse Elenga, Principal Investigator — CHG Andrée Rosemon Cayenne; Natacha Entz Werle, Principal Investigator — Hautepierre Strasbourg; Thomas Girard, Principal Investigator — Hotel Dieu Paris; Martine Levine, Principal Investigator — Robert Debré Paris; Benoit Martha, Principal Investigator — CH Chalon sur Soane; Sandrine Anne Martha, Principal Investigator — Chalon sur Saone; Patrice Poubeau, Principal Investigator — CHR Réunion St Pierre; Jean Marc Treluyer, Principal Investigator — CIC Necker Paris; Louis Bernard, Principal Investigator — Hôpital Bretonneau Tours; Michel Dupon, Principal Investigator — Hôpital Pellegrin Bordeaux; David Zucman, Principal Investigator — Hôpital Foch Suresnes; Anne Simon, Principal Investigator — Pitié Salpétrière Paris; Isabellle Poizot Martin, Principal Investigator — Ste Marguerite Marseille; Thierry Prazuck, Principal Investigator — CHR Orléans; Eric Doré, Principal Investigator — CHU Estains Clermont Ferrand; Catherine Gaud, Principal Investigator — CHR Site Felix Guyon Bellepierre La Réunion
Locations (1):
- Hôpitaux (voir liste jointe), De France, France

REFERENCES:
- See also: Related Info — http://anrs.fr